CLINICAL TRIAL: NCT01194505
Title: Comparison of Posterior Lumbar Plexus Block Plus Sciatic Nerve Block With Sciatic Plus Femoral Plus Obturator Nerve Block for Anterior Cruciate Ligament Reconstruction
Brief Title: Ultrasound Guided Obturator Nerve Block for Anterior Cruciate Ligament Reconstruction (ACL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Metaxia Bareka, Anesthesiologist, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ACLObturator
Record Dates: First submitted 2010-09-01; First posted 2010-09-03 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Anterior Cruciate Ligament; Surgery
Keywords: anterior cruciate ligament reconstruction; obturator nerve block; sciatic nerve block; femoral nerve block; posterior lumbar plexus block; ultrasound guided nerve block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient, the orphopaedic surgeon and the anesthesiologist in the OR did not know at which group the patient belonged to.
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACL, sciatic, femoral, obturator (Active Comparator): ACL reconstruction surgery under ultrasound guided sciatic nerve block plus femoral nerve block plus obturator nerve block
  Interventions: Other: Sciatic, femoral, obturator nerve blocks
- ACL, sciatic nerve block, posterior lumbar plexus block (Active Comparator): ACL reconstruction surgery under ultrasound guided sciatic nerve block plus posterior lumbar plexus block
  Interventions: Other: Sciatic nerve block, posterior lumbar plexus block

INTERVENTIONS:
Other: Sciatic, femoral, obturator nerve blocks — Ultrasound guided blocks with ropivacaine
  Arms: ACL, sciatic, femoral, obturator
Other: Sciatic nerve block, posterior lumbar plexus block — Ultrasound and neurostimulator nerve blocks with ropivacaine
  Arms: ACL, sciatic nerve block, posterior lumbar plexus block

SUMMARY:
Anterior Cruciate Ligament ACL reconstruction can be performed under the combination of posterior lumbar plexus block plus sciatic nerve block. The investigators can have the same outcome by performing instead of posterior lumbar plexus block more peripheral nerve blocks. More specifically under the combination of sciatic nerve block plus femoral nerve block plus obturator nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years old
* ASA I - II
* ACL reconstruction surgery

Exclusion Criteria:

* Coagulopathy disorders
* Infection at the puncture site for the interscalene block
* Neurologic deficit in the arm that is going to be operated
* Allergy to local anesthetics
* BMI > 35
* Psychiatric disorders
* Patient's refusal
* Problems with patient communication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of ACL reconstruction surgery under ultrasound guided sciatic nerve block plus femoral nerve block plus obturator nerve block measured with Pain Score on the Visual Analog Scale | 45 min
  If the patient complains for pain > 4 in VAS and there is no relief with fentanyl administration the anesthesia plan converts to general anesthesia with laryngeal mask

SECONDARY OUTCOMES:
Intraoperative opioid consumption for ACL reconstruction surgery under ultrasound guided sciatic nerve block plus femoral nerve block plus obturator nerve block | Intraoperatively
Postoperative opioid consumption for ACL reconstruction surgery under ultrasound guided sciatic nerve block plus femoral nerve block plus obturator nerve block | 24h

CONTACTS AND LOCATIONS:
Overall Officials: Metaxia Bareka, Medicine, Principal Investigator — Larissa University Hospital; George Vretzakis, Medicine, Study Director — Larissa University Hospital; Eleni Chantzi, Medicine, Study Chair — Larissa University Hospital; Michael Hantes, Medicine, Study Chair — Larissa University Hospital; Eleni Askitopoulou, Medicine, Study Chair — Heraklion University Hospital; Marina Simaioforidou, Medicine, Study Chair — Larissa University Hospital
Locations (1):
- Larissa University Hospital, Larissa, Thessaly, Greece

REFERENCES:
- [Background] Zwissler B. [An exceptional author and publisher is leaving : Retirement of Reinhard Larsen from the editorial board of Der Anaesthesist]. Anaesthesist. 2010 Jan;59(1):5-6. doi: 10.1007/s00101-009-1649-2. No abstract available. German. PMID 20094695
- [Background] Enneking FK, Chan V, Greger J, Hadzic A, Lang SA, Horlocker TT. Lower-extremity peripheral nerve blockade: essentials of our current understanding. Reg Anesth Pain Med. 2005 Jan-Feb;30(1):4-35. doi: 10.1016/j.rapm.2004.10.002. No abstract available. PMID 15690265
- [Background] Fanelli G, Casati A, Aldegheri G, Beccaria P, Berti M, Leoni A, Torri G. Cardiovascular effects of two different regional anaesthetic techniques for unilateral leg surgery. Acta Anaesthesiol Scand. 1998 Jan;42(1):80-4. doi: 10.1111/j.1399-6576.1998.tb05084.x. PMID 9527749
- [Background] Hadzic A, Karaca PE, Hobeika P, Unis G, Dermksian J, Yufa M, Claudio R, Vloka JD, Santos AC, Thys DM. Peripheral nerve blocks result in superior recovery profile compared with general anesthesia in outpatient knee arthroscopy. Anesth Analg. 2005 Apr;100(4):976-981. doi: 10.1213/01.ANE.0000150944.95158.B9. PMID 15781509
- [Background] Jankowski CJ, Hebl JR, Stuart MJ, Rock MG, Pagnano MW, Beighley CM, Schroeder DR, Horlocker TT. A comparison of psoas compartment block and spinal and general anesthesia for outpatient knee arthroscopy. Anesth Analg. 2003 Oct;97(4):1003-1009. doi: 10.1213/01.ANE.0000081798.89853.E7. PMID 14500148
- [Background] Morin AM, Pandurovic M, Eberhart LH, Wagner S, Kunz C, Nussle W, Geiger P, Mehrkens HH. [Is a blockade of the lateral cutaneous nerve of the thigh an alternative to the classical femoral nerve blockade for knee joint arthroscopy? A randomised controlled study]. Anaesthesist. 2005 Oct;54(10):991-9. doi: 10.1007/s00101-005-0879-1. German. PMID 15968551
- [Background] Heller AR, Fuchs A, Rossel T, Vicent O, Wiessner D, Funk RH, Koch T, Litz RJ. Precision of traditional approaches for lumbar plexus block: impact and management of interindividual anatomic variability. Anesthesiology. 2009 Sep;111(3):525-32. doi: 10.1097/ALN.0b013e3181af64b6. PMID 19672183
- [Background] Winnie AP, Ramamurthy S, Durrani Z. The inguinal paravascular technic of lumbar plexus anesthesia: the "3-in-1 block". Anesth Analg. 1973 Nov-Dec;52(6):989-96. No abstract available. PMID 4796576
- [Background] Kessler J, Marhofer P, Rapp HJ, Hollmann MW. [Ultrasound-guided anaesthesia of peripheral nerves. The new challenge for anaesthesiologists]. Anaesthesist. 2007 Jul;56(7):642-55. doi: 10.1007/s00101-007-1223-8. German. PMID 17576526
- [Background] Danelli G, Ghisi D, Fanelli A, Ortu A, Moschini E, Berti M, Ziegler S, Fanelli G. The effects of ultrasound guidance and neurostimulation on the minimum effective anesthetic volume of mepivacaine 1.5% required to block the sciatic nerve using the subgluteal approach. Anesth Analg. 2009 Nov;109(5):1674-8. doi: 10.1213/ANE.0b013e3181b92372. PMID 19843807
- [Background] Klein SM, Evans H, Nielsen KC, Tucker MS, Warner DS, Steele SM. Peripheral nerve block techniques for ambulatory surgery. Anesth Analg. 2005 Dec;101(6):1663-1676. doi: 10.1213/01.ANE.0000184187.02887.24. PMID 16301239
- [Background] Greengrass RA, Klein SM, D'Ercole FJ, Gleason DG, Shimer CL, Steele SM. Lumbar plexus and sciatic nerve block for knee arthroplasty: comparison of ropivacaine and bupivacaine. Can J Anaesth. 1998 Nov;45(11):1094-6. doi: 10.1007/BF03012398. PMID 10021959
- [Background] Freeman MA, Wyke B. The innervation of the knee joint. An anatomical and histological study in the cat. J Anat. 1967 Jun;101(Pt 3):505-32. No abstract available. PMID 6051731
- [Background] Boezaart A. Continuous femoral Nerve Block for Pain Management in Total Knee Arthoplasty. AAOS, Orthopaedic Knowledge On Line
- [Background] Simeoforidou M, Bareka M, Basdekis G, Tsiaka K, Chantzi E, Vretzakis G. Peripheral nerve blockade as an exclusive approach to obturator nerve block in anterior cruciate ligament reconstructive surgery. Korean J Anesthesiol. 2013 Nov;65(5):410-7. doi: 10.4097/kjae.2013.65.5.410. Epub 2013 Nov 29. PMID 24363843
- [Background] Bareka M, Hantes M, Arnaoutoglou E, Vretzakis G. Superior perioperative analgesia with combined femoral-obturator-sciatic nerve block in comparison with posterior lumbar plexus and sciatic nerve block for ACL reconstructive surgery. Knee Surg Sports Traumatol Arthrosc. 2018 Feb;26(2):478-484. doi: 10.1007/s00167-017-4525-7. Epub 2017 Mar 18. PMID 28315922